CLINICAL TRIAL: NCT05659654
Title: A Single-center, Open, Single-arm Clinical Study on the Application of Ursodeoxycholic Acid for the Prevention of SARS-CoV-2 Infections
Brief Title: The Application of Ursodeoxycholic Acid for the Prevention of SARS-CoV-2 Infection (COVID-19)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: QTJC2022056
Record Dates: First submitted 2022-12-18; First posted 2022-12-21 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2023-03

CONDITIONS: COVID-19
Keywords: ursodeoxycholic acid; COVID-19; prevention
MeSH Terms: conditions — COVID-19 | interventions — Ursodeoxycholic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Take ursodeoxycholic acid capsules daily for 4 weeks from the date of enrollment (Experimental): Healthy volunteers took ursodeoxycholic acid capsules daily for 4 weeks from the date of enrollment
  Interventions: Drug: Ursodeoxycholic acid

INTERVENTIONS:
Drug: Ursodeoxycholic acid — 250 mg/capsule, 2 capsules per day, for 4 weeks

SUMMARY:
Evaluation of the efficacy and safety of ursodeoxycholic acid in blocking the transmission of infectious novel coronaviruses in a population of medical workers

DETAILED DESCRIPTION:
This is a single-center, open-ended, single-arm clinical study to evaluate the effectiveness of daily ursodeoxycholic acid plus routine protective measures for the prevention of novel coronavirus infection. The target sample size is 130 medical workers and each healthy volunteer will be followed weekly for nucleic acid/antigen testing or disease progression over an 8-week period for new crown infections.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 - 65 years old.
2. No restriction on gender.
3. Medical-related personnel (working hours >20 hours per week) serving during the COVID-19 outbreak, including physicians, nurses, medical technicians, administrators, and medical students
4. COVID-19 nucleic acid test negative within 48 hours
5. Sign the informed consent form

Exclusion Criteria:

1. Exhibit COVID-19 symptoms, including fever, muscle pain, headache, cough, sore throat, and loss of smell and taste
2. Previous infection with novel coronavirus within 6 months
3. Previous (past 30 days), current or planned (during the study period) use of immunomodulatory-related drugs
4. Those with allergy or intolerance to ursodeoxycholic acid, gallbladder or bile duct disease, severe liver failure, or liver function impairment
5. Pregnancy and lactation
6. Use of drugs with which ursodeoxycholic acid is contraindicated
7. Other reported health conditions that make participation in the study not in the best interest of the individual

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2022-12-16 (Actual); Primary Completion 2023-03-03 (Actual); Study Completion 2023-03-08 (Actual)

PRIMARY OUTCOMES:
Prevalence of novel coronavirus infection | Receiving 4 weeks of continuous ursodeoxycholic acid
  Prevalence of novel coronavirus infection in healthy volunteers receiving 4 weeks of continuous ursodeoxycholic acid plus conventional protection during the study period

SECONDARY OUTCOMES:
The proportion of people infected with novel coronavirus who turned severe | 8 weeks
  The proportion of people infected with novel coronavirus who turned severe
The number of days that symptoms of a novel coronavirus infection,muscle aches persisted in the population infected with novel coronavirus | 8 weeks
  The number of days that symptoms of a novel coronavirus infection such as fever, sore throat, headache, and muscle aches persisted in the population infected with novel coronavirus, and the number of days that the nucleic acid/antigen turned negative.
The rate of positive serological antibodies in the population of healthy volunteers | 8 weeks
  The rate of positive serological antibodies in the population of healthy volunteers
The incidence of adverse events | 8 weeks
  The incidence of adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese Academy of Medical Science and Blood Disease Hospital,CAMS & PUMC, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Yes

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2023-03-06): https://cdn.clinicaltrials.gov/large-docs/54/NCT05659654/Prot_ICF_001.pdf